CLINICAL TRIAL: NCT01184664
Title: Effects of a Combination of Varenicline and Transdermal Nicotine Patch on Post-quitting Urges to Smoke
Brief Title: Combination of Nicotine Replacement Therapy (NRT) and Varenicline to Increase Cessation of Tobacco (CONVICT Study)
Acronym: CONVICT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Professor Peter Hajek, Professor of Clinical Psychology, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: qmul250510; 2010-022334-92 (EudraCT Number)
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Tobacco Dependence; Smoking Cessation
Keywords: Smoking cessation; Tobacco dependence; Varenicline; Nicotine Replacement Therapy; Combination therapy
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Tobacco Use Cessation Devices; Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline + Active Patch (Experimental): Participants will use varenicline (1mg BD) + an active, 15mg/16hr Nicotine Patch
  Interventions: Drug: Nicotine Patch; Drug: Varenicline
- Varenicline + Placebo Patch (Placebo Comparator): Participants will use varenicline (1mg BD) + a Placebo Nicotine Patch
  Interventions: Drug: Placebo; Drug: Varenicline

INTERVENTIONS:
Drug: Nicotine Patch — Varenicline + nicotine patch
  Other Names: Champix; Chantix
  Arms: Varenicline + Active Patch
Drug: Placebo — Varenicline + placebo patch
  Other Names: Champix; Chantix
  Arms: Varenicline + Placebo Patch
Drug: Varenicline — All participants will receive a standard dose of varenicline (12 weeks).
  Other Names: Champix; Chantix

SUMMARY:
Varenicline and nicotine replacement therapy (NRT) are both effective smoking cessation treatments. Anecdotally smokers who are finding their quit attempt difficult have reported benefiting from adding NRT to varenicline. This proof-of-principle placebo-controlled double-blind study will examine whether combining NRT and varenicline provides better withdrawal and craving relief than varenicline alone. A total of 120 smokers would be randomised to receive varenicline +15mg/16hr patch or varenicline + placebo patch. All participants will receive standard NHS Stop Smoking Service support. The primary outcome would be ratings of craving and withdrawal discomfort 24 hours and one week after the target quit date.

ELIGIBILITY:
Inclusion Criteria:

* Smokers seeking treatment
* Aged 18 and over
* Consenting to take part in the trial

Exclusion Criteria:

* Pregnant or breastfeeding
* End-stage renal disease
* Unable to fill in questionnaires in English
* Previous allergy to Varenicline
* Previous allergy to Nicotine Patches Previous allergy to varenicline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Rating of urges to smoke one week after the target quit date assessed by Mood and Physical Symptoms Scale | 1 week
  Rating of urges to smoke will be assessed using the Mood and Physical Symptoms Scale

SECONDARY OUTCOMES:
Validated abstinence rates over weeks 1-12 post target quit date | 12 weeks post target quit date
Rating of withdrawal symptoms up to 4-weeks post quitting assessed by Mood and Physical Symptoms Scale | 4-weeks post quitting
Profile of all adverse effects reported up to 12-weeks post quitting | Up to 12-weeks post quitting
Ratings of urges to smoke 24 hours after the target quit date | 24 hours
  Urges to smoke at 24 hours after the target quit date will be assessed using the Mood & Physical Symptoms Scale

CONTACTS AND LOCATIONS:
Overall Officials: Al-Rehan A A Dhanji, MB BS BSc MRCS, Principal Investigator — Queen Mary University of London
Locations (2):
- United Kingdom (2):
  - Tobacco Dependence Research and Treatment Unit, London
  - Tobacco Dependence Research Unit, London

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Hajek P, Smith KM, Dhanji AR, McRobbie H. Is a combination of varenicline and nicotine patch more effective in helping smokers quit than varenicline alone? A randomised controlled trial. BMC Med. 2013 May 29;11:140. doi: 10.1186/1741-7015-11-140. PMID 23718718